

Study Code: UDDGait SAP Version: 1.0

Date: February 4th, 2020

# **Statistical Analysis Plan**

| Study Code: | UDDGait |
|----------------------------|----------------------|
| Study Title: | UDDGait paper III |
| Biostatistician: | Lars Berglund |
| Data Manager: | Vilmantas Giedraitis |
| Project Leader: | Anna Cristina Åberg |
| SAP version: | 1.0 |
| Changes from last version: | N/A |



Study Code: UDDGait SAP Version: 1.0

Date: February 4th, 2020

## **Table of Contents**

| Introduction | 3 |
|-------------------------------------------|---|
| Abbreviations and Variable List | |
| Abbreviations | |
| Variable List | 4 |
| Study Objectives and Endpoints | |
| Objectives | |
| Primary Objectives | 4 |
| Endpoint | |
| Primary Endpoint | 5 |
| Study Design | |
| Definition of Analysis Population | 5 |
| Statistical Description and Analysis | 5 |
| Derived variables | 5 |
| Baseline Characteristics | 5 |
| Primary Analyses | 6 |
| Estimated Effects | |
| Logistic Regression Models | |
| Receiving Operator Characteristics Curves | |
| Output Shell | |
| References | 7 |



Study Code: UDDGait Date: February 4th, 2020

SAP Version: 1.0

#### Introduction

The present statistical analysis plan (SAP) outlines statistical description and analysis for paper III from the UDDGait study (1). The paper will present data from the baseline and the follow-up at two years after baseline for patients with subjective cognitive impairment (SCI) or mild cognitive impairment (MCI) at baseline. Results will be compiled into a statistical report for which the output tables and figures are displayed in Table 3.

### **Abbreviations and Variable List**

#### **Abbreviations**

CDT Clock Drawing Test

UDDGait Uppsala-Dalarna Dementia and Gait study

MCI Mild Cognitive Impairment

MMSE Mini Mental State Examination

SAP Statistical Analysis Plan

SCI Subjective Cognitive Impairment

TUG Timed Up and Go test



Study Code: UDDGait Date: February 4th, 2020

SAP Version: 1.0

#### Variable List

Table 1. Variable list (all variables measured at baseline if not otherwise stated)

| Variable (unit) | Variable | Variable | SAS name |
|---|---|---|---|
| | scale <sup>1</sup> | rôle | |
| Age (years) | С | Confounder | D005 |
| Age group (<72 years/>=72 years) | D | Strata | AGEGR |
| Gender | D | Confounder | D006 |
| Education (high/low) | D | Confounder | D008 |
| Diagnoses at two years (dementia/non-dementia) | D | Outcome | F10C |
| MMSE | С | Confounder | D041 |
| TUG single task, s | С | Predictor | D021 |
| TUG dual task animals, s | С | Predictor | D023 |
| TUG dual task animals, number of correct animals | С | Predictor | D024 |
| TUG dual task cost animals, % | С | Predictor | D023C |
| TUG dual task animals, number of animals per 10s | С | Predictor | D023S |
| TUG dual task months, s | С | Predictor | D027 |
| TUG dual task animals, number of correct months | С | Predictor | D028 |
| TUG dual task costs months, % | С | Predictor | D027C |
| TUG dual task months, number of months per 10s | С | Predictor | D027S |
| Diagnoses (SCI/MCI) | D | | D10GR4 |
| Marital status | D | | D007 |
| CDT | С | | D042 |
| Word flow | С | | D043 |
| Bohannon's balance test | С | | D050 |
| Depression scale | С | | D046 |
| Height | С | | D011 |
| TMT A | D | | D044 |
| TMT B | D | | D045 |
| GMF help | С | | D047 |
| GMF pain | С | | D048 |
| GMF anxiety | С | | D049 |
| Hand grip | С | | D051 |

<sup>&</sup>lt;sup>1</sup>C = continuous variable, D = dichotomous variable.

## **Study Objectives and Endpoints**

### **Objectives**

### **Primary Objectives**

The primary objective is to investigate if dual task variables are associated with incident dementia from baseline to follow-up after two years for patients with subjective cognitive impairment (SCI) or mild cognitive impairment (MCI) at baseline, unadjusted and adjusted for age, gender, education level and Mini Mental State Examination (MMSE). Further, this objective will be examined in younger (< 72 years) and older (>= 72 years) patients.



Study Code: UDDGait Date: February 4th, 2020

SAP Version: 1.0

### **Endpoint**

### **Primary Endpoint**

The primary endpoint is the dichotomous variable diagnoses of dementia vs. non-dementia at the two years follow-up.

## **Study Design**

The study design is prospective longitudinal.

## **Definition of Analysis Population**

The study population to be analysed consists of the study patients with diagnoses SCI or MCI at baseline and for whom a dementia diagnosis could be determined at two years after baseline.

## **Statistical Description and Analysis**

#### Derived variables

The measures "animals/10 s" and "months/10 s" were calculated as 10\*(TUGdt number of words/TUGdt time score). Dual-task cost, i.e. the relative time difference between TUGst and TUGdt, was calculated as 100\*(TUGdt time score –TUGst time score)/TUGst time score.

#### **Baseline Characteristics**

All baseline variables in Table 1 will be summarized for the whole study population and by incident dementia (yes/no) at two years follow-up. Further, all baseline variables in Table 1 will be summarized by younger (< 72 years) and older (>= 72 years) patients for the whole age stratum and by incident dementia (yes/no) at two years follow-up. The continuous variables will be described with number of observations, number of missing observations, mean, standard deviation, median and minimum and maximum values. Dichotomous and categorical variables will be described with numbers, number of missing observations, and percentages.



Study Code: UDDGait Date: February 4th, 2020

SAP Version: 1.0

### **Primary Analyses**

All statistical tests and confidence intervals are two-sided (where applicable) and the region p < 0.05 is used to declare a statistically significant result. No adjustments for multiple tests will be made. No imputations of missing data will be made.

#### **Estimated Effects**

The aims of the analyses of the primary and secondary endpoints will be investigated with estimated logistic regression models. The results from the models will be presented, for each continuous predictor, as estimated odds ratios, with 95 % confidence intervals, of a one standard deviation impaired change of the predictor, and a p value for test of the null hypothesis that the true odds ratio is unity. Impaired changes imply that for the time scores of TUG single task, s, TUG dual task animals, s TUG dual task months, s as well as TUG dual task cost animals, %, and TUG dual task cost months, %, the ORs express the risk increase per one standard deviation *increase* of the variable. Whereas for the number of animals and number of months, as well as "animals/10 s" and "months/10 s" the ORs express the risk increase per one standard deviation *decrease* of the variable.

Logistic regressions will be estimated univariate for each TUG variable and with adjustment for age, gender, education and MMSE.

### **Logistic Regression Models**

The logistic regression models to be estimated are shown in Table 2.

Table 2. Logistic regression models

| Objective | Outcome(s) | Predictors |
|---|---|---|
| Primary | Incident dementia | Each dual task predictor individually |
| Primary | Incident dementia | Each dual task predictor individually, and age, gender, education and MMSE |
| Primary | Incident dementia | Each dual task predictor individually stratified by age groups < 72 years and >= 72 years |
| Primary | Incident dementia | Each dual task predictor individually<br>and age, gender, education and MMSE<br>stratified by age groups < 72 years and<br>>= 72 years |



Study Code: UDDGait Date: February 4th, 2020

SAP Version: 1.0

### **Receiving Operator Characteristics Curves**

Results from the models will be presented with estimated effects and 95 % confidence intervals and p values.

Predictive capacity for each TUG variable will be illustrated with receiving operator characteristics (ROC) curves and c statistics (areas under ROC curves). These curves will be presented univariate and with the incremental effect of the TUG variable over a model with age, gender, education and MMSE.

The above described analyses will also be presented stratified by age groups < 72 years and >= 72 years.

### **Output Shell**

In the following table the names and contents of output tables and figures are displayed.

Table 3. Output shell

| Table | Content |
|---|---|
| Table 1a | Descriptive table for all variables, in total and by incident dementia (yes/no) |
| Table 1b | Descriptive table for all variables, in total and by incident dementia (yes/no) stratified by age groups < 72 years and >= 72 years |
| Table 2 | Results of logistic regression models in SAP Table 2 |
| Figure 1.1-1.9 | ROC curve for each TUG variable |
| Figure 2.2-2.9 | ROC curve for the incremental predictive capacity for each TUG variable over the model with age, gender, education and MMSE |
| Figure 3.1-3.9 | ROC curve for each TUG variable stratified by age groups < 72 years and >= 72 years |
| Figure 4.1-4.9 | ROC curve for the incremental predictive capacity for each TUG variable over the model with age, gender, education and MMSE stratified by age groups < 72 years and >= 72 years |

## References

1. Project plan UDDGait



Study Code: UDDGait SAP Version: 1.0

Date: February 4th, 2020